CLINICAL TRIAL: NCT01541020
Title: Inspiratory Resistive Loading and Proprioceptive Postural Control in Healthy Individuals and Individuals With Recurrent Low Back Pain
Brief Title: Inspiratory Resistive Loading and Proprioceptive Postural Control
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Prof. dr. Simon Brumagne, KU Leuven
Other Study IDs: 2011_SBrumagne_HealthyLBP; 1.5.104.03, G.0674.09 (Other Grant/Funding Number: Research Foundation Flanders (FWO))
Record Dates: First submitted 2012-01-04; First posted 2012-02-29 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2012-01

CONDITIONS: Low Back Pain; Respiratory Loading; Proprioceptive Impairment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy individuals
- Individuals with low back pain

SUMMARY:
Proprioceptive weighting changes may explain differences in postural control performance. In addition, the respiratory movement has a disturbing effect on postural balance. Postural balance seems to be impaired in individuals with respiratory disorders. Besides the essential role of respiration, the diaphragm may also play an important role in the control of the trunk and postural balance. Deficits in proprioception are found in a subgroup of patients with low back pain. In addition, disorders of respiration have been identified as strongly related to low back pain.

The aim of the study is to clarify whether loading of the inspiratory muscles has a negative effect upon proprioceptive postural control in healthy individuals and individuals with recurrent low back pain.

ELIGIBILITY:
Inclusion Criteria individuals with low back pain:

* Age: 18-45 years old
* At least 1 year of low back pain with/without referred pain in buttock/thigh
* At least 3 episodes of disabling low back pain
* At least a score of 20% on the Oswestry Disability Index
* Willingness to sign the informed consent

Inclusion Criteria healthy individuals:

* Age: 18-45 years old
* No history of low back pain
* A score of 0% on the Oswestry Disability Index
* Willingness to sign the informed consent

Exclusion Criteria:

* History of major trauma and/or major orthopedic surgery of the spine, the pelvis or the lower quadrant
* One of the following conditions: Parkinson, multiple sclerosis, stroke, history of vestibular disorder, respiratory disease, pregnancy
* Radicular symptoms
* Not Dutch-speaking
* Strong opioids
* Neck pain
* Smoking history

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young flemish volunteers
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proprioceptive postural control | 1 year
  Center of pressure displacement (force plate) in standing in response to local muscle vibration on ankle and back muscles to specifically detect the role of proprioception in postural control.

SECONDARY OUTCOMES:
Back muscle oxygenation | 1 year
  Near infrared spectroscopy: tissue oxygenation index (TOI) and haemoglobin
Kinematics | 1 year
  piezoresistive accelerometers
Respiratory muscle force | 1 year
  maximal inspiratory pressure - maximal expiratory pressure

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brumagne, PhD, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Janssens L, Brumagne S, Polspoel K, Troosters T, McConnell A. The effect of inspiratory muscles fatigue on postural control in people with and without recurrent low back pain. Spine (Phila Pa 1976). 2010 May 1;35(10):1088-94. doi: 10.1097/BRS.0b013e3181bee5c3. PMID 20393397